CLINICAL TRIAL: NCT05874635
Title: Use of Signos mHealth Platform in Participants With Non-Insulin Dependent Type 2 Diabetes: Weight and Blood Glucose
Brief Title: Signos DM2 Empowerment Study (SIGNOS-CGM-EMPOWER-201-2022)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Signos Inc (Industry)
Responsible Party: Principal Investigator, Stephanie Kim, M.D., MPH, Principal Investigator, Signos Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201-2022
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Weight Loss; Metabolic Syndrome; Diabetes Mellitus, Type 2; Central Obesity; Insulin Resistance; Glucose Intolerance; Metabolic Glucose Disorders
Keywords: health and wellness; excess adiposity
MeSH Terms: conditions — Weight Loss; Metabolic Syndrome; Diabetes Mellitus, Type 2; Obesity, Abdominal; Insulin Resistance; Glucose Intolerance; Glucose Metabolism Disorders

STUDY DESIGN:
Intervention Model Description: Open label single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Signos digital health app and CGM (Experimental): For all consented participants, the Signos app will use CGM data to provide recommendations customized to users for promoting general health and wellness.
  Interventions: Device: Continuous Glucose Monitor Device

INTERVENTIONS:
Device: Continuous Glucose Monitor Device — Continuous glucose monitoring automatically tracks blood glucose levels, also called blood sugar, throughout the day and night. You can see your glucose level anytime at a glance. You can also review how your glucose changes over a few hours or days to see trends. Seeing glucose levels in real time can help you make more informed decisions throughout the day about how to balance your food and physical activity.
  Other Names: CGM

SUMMARY:
The use of continuous glucose monitoring (CGM) in earlier data has inspired behavioral changes leading to improved adherence to an exercise plan in individuals and eating habits in people with diabetes. Mobile health (mHealth) platforms provide satisfactory, easy-to-use tools to help participants in the pursuit of weight change goals. We hypothesize that the use of CGM data and the Signos mHealth platform will assist with weight control in a population of people with type 2 diabetes mellitus who are not using insulin.

DETAILED DESCRIPTION:
The scope of this study is to enroll existing and new Signos non-insulin dependent type 2 diabetes mellitus users in a volunteer study that utilizes a continuous glucose monitor (CGM) and mobile health application [Signos] to optimize general wellness and body weight and composition. This is a no more than minimal risk study.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of Type 2 Diabetes; determined by review of subject-provided most recent Hg A1c.
* Subject is under current care of a primary care provider or specialist
* Clearance by medical provider to participate in diet, physical activity, and lifestyle changes
* 18 years and above
* Own a smartphone and be willing to install the Signos App to personally receive text messages or have access to a web-based survey to self-report their weight.
* Willingness to complete quality of life questionnaires or other in-app surveys.
* Willingness to use CGM device
* Able to speak and read English
* Be a Signos mHealth (mobile/web-based) user

Exclusion Criteria:

* Medical diagnosis of Type 1 Diabetes
* Type 2 Diabetes currently using insulin or most recent A1c ≥10%
* Severe hypoglycemia <54 mg/dl resulting in seizure or unconsciousness, or requiring assistance/EMS/hospitalization - within 3 months prior to enrollment
* Current medical diagnosis of an eating disorder (such as anorexia nervosa or bulimia)
* Medical conditions (e.g., such as seizure disorder) requiring a specific medical diet.
* Inborn error of metabolism such as phenylketonuria (PKU), glycogen storage disease, fructose intolerance, Maple Sugar Urine Disease (MSUD).
* History of 10 or more soft tissue skin infections (such as cellulitis or abscesses)
* Intolerable skin reaction from adhesive
* Currently taking any of the following medications: Clozapine, Hydroxyurea, or any form of insulin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2028-05-10 (Estimated); Study Completion 2029-05-10 (Estimated)

PRIMARY OUTCOMES:
Glucose Metrics via Continuous Glucose Measurement (CGM) | During enrollment in the trial for a maximum of 5 years, including a 1 year follow up period, for a maximum of 6 years.
  Glucose measured in mg/dl
Change in weight in pounds | During enrollment in the trial for a maximum of 5 years, including a 1 year follow up period, for a maximum of 6 years.
  Change in number of pounds
App engagement | During enrollment in the trial for a maximum of 5 years, including a 1 year follow up period, for a maximum of 6 years.
  Meals logged, Exercises logged, Activities completed

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Kim, MD, Principal Investigator — Signos Inc
Locations (1):
- Signos, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hall H, Perelman D, Breschi A, Limcaoco P, Kellogg R, McLaughlin T, Snyder M. Glucotypes reveal new patterns of glucose dysregulation. PLoS Biol. 2018 Jul 24;16(7):e2005143. doi: 10.1371/journal.pbio.2005143. eCollection 2018 Jul. PMID 30040822
- [Result] Adams OP. The impact of brief high-intensity exercise on blood glucose levels. Diabetes Metab Syndr Obes. 2013;6:113-22. doi: 10.2147/DMSO.S29222. Epub 2013 Feb 27. PMID 23467903
- [Result] Zeevi D, Korem T, Zmora N, Israeli D, Rothschild D, Weinberger A, Ben-Yacov O, Lador D, Avnit-Sagi T, Lotan-Pompan M, Suez J, Mahdi JA, Matot E, Malka G, Kosower N, Rein M, Zilberman-Schapira G, Dohnalova L, Pevsner-Fischer M, Bikovsky R, Halpern Z, Elinav E, Segal E. Personalized Nutrition by Prediction of Glycemic Responses. Cell. 2015 Nov 19;163(5):1079-1094. doi: 10.1016/j.cell.2015.11.001. PMID 26590418
- [Result] Baron AD. Impaired glucose tolerance as a disease. Am J Cardiol. 2001 Sep 20;88(6A):16H-9H. doi: 10.1016/s0002-9149(01)01832-x. PMID 11576521
- [Result] Brown A, McArdle P, Taplin J, Unwin D, Unwin J, Deakin T, Wheatley S, Murdoch C, Malhotra A, Mellor D. Dietary strategies for remission of type 2 diabetes: A narrative review. J Hum Nutr Diet. 2022 Feb;35(1):165-178. doi: 10.1111/jhn.12938. Epub 2021 Sep 1. PMID 34323335
- [Result] Chin SO, Keum C, Woo J, Park J, Choi HJ, Woo JT, Rhee SY. Successful weight reduction and maintenance by using a smartphone application in those with overweight and obesity. Sci Rep. 2016 Nov 7;6:34563. doi: 10.1038/srep34563. PMID 27819345
- [Result] Ebbeling CB, Knapp A, Johnson A, Wong JMW, Greco KF, Ma C, Mora S, Ludwig DS. Effects of a low-carbohydrate diet on insulin-resistant dyslipoproteinemia-a randomized controlled feeding trial. Am J Clin Nutr. 2022 Jan 11;115(1):154-162. doi: 10.1093/ajcn/nqab287. PMID 34582545
- [Result] Ehrhardt N, Al Zaghal E. Behavior Modification in Prediabetes and Diabetes: Potential Use of Real-Time Continuous Glucose Monitoring. J Diabetes Sci Technol. 2019 Mar;13(2):271-275. doi: 10.1177/1932296818790994. Epub 2018 Aug 1. PMID 30066574
- [Result] The Lancet Diabetes Endocrinology. Metabolic health: a priority for the post-pandemic era. Lancet Diabetes Endocrinol. 2021 Apr;9(4):189. doi: 10.1016/S2213-8587(21)00058-9. Epub 2021 Mar 4. No abstract available. PMID 33676599
- [Result] Galderisi A, Giannini C, Weiss R, Kim G, Shabanova V, Santoro N, Pierpont B, Savoye M, Caprio S. Trajectories of changes in glucose tolerance in a multiethnic cohort of obese youths: an observational prospective analysis. Lancet Child Adolesc Health. 2018 Oct;2(10):726-735. doi: 10.1016/S2352-4642(18)30235-9. Epub 2018 Aug 24. PMID 30236381
- [Result] Gonzalez-Rodriguez M, Pazos-Couselo M, Garcia-Lopez JM, Rodriguez-Segade S, Rodriguez-Garcia J, Tunez-Bastida C, Gude F. Postprandial glycemic response in a non-diabetic adult population: the effect of nutrients is different between men and women. Nutr Metab (Lond). 2019 Jul 17;16:46. doi: 10.1186/s12986-019-0368-1. eCollection 2019. PMID 31346341
- [Result] Guyenet SJ, Schwartz MW. Clinical review: Regulation of food intake, energy balance, and body fat mass: implications for the pathogenesis and treatment of obesity. J Clin Endocrinol Metab. 2012 Mar;97(3):745-55. doi: 10.1210/jc.2011-2525. Epub 2012 Jan 11. PMID 22238401
- [Result] Hamley S, Kloosterman D, Duthie T, Dalla Man C, Visentin R, Mason SA, Ang T, Selathurai A, Kaur G, Morales-Scholz MG, Howlett KF, Kowalski GM, Shaw CS, Bruce CR. Mechanisms of hyperinsulinaemia in apparently healthy non-obese young adults: role of insulin secretion, clearance and action and associations with plasma amino acids. Diabetologia. 2019 Dec;62(12):2310-2324. doi: 10.1007/s00125-019-04990-y. Epub 2019 Sep 6. PMID 31489455
- [Result] Hyde PN, Sapper TN, Crabtree CD, LaFountain RA, Bowling ML, Buga A, Fell B, McSwiney FT, Dickerson RM, Miller VJ, Scandling D, Simonetti OP, Phinney SD, Kraemer WJ, King SA, Krauss RM, Volek JS. Dietary carbohydrate restriction improves metabolic syndrome independent of weight loss. JCI Insight. 2019 Jun 20;4(12):e128308. doi: 10.1172/jci.insight.128308. eCollection 2019 Jun 20. PMID 31217353